CLINICAL TRIAL: NCT06610708
Title: Pre-Intervention Rehabilitation to Optimize Patient Selection for Chronic Total Occlusion Percutaneous Coronary Interventions (PREHAB-CTO Study)
Brief Title: Feasibility of a Cardiac Rehabilitation Program for CTO Patients Before PCI Treatment
Acronym: PREHAB-CTO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Luiz Ybarra (Other)
Collaborators: Academic Medical Organization of Southwestern Ontario (Other); University of Western Ontario, Canada (Other)
Responsible Party: Sponsor-Investigator, Luiz Ybarra, Interventional Cardiologist, Principal Investigator, London Health Sciences Centre
Organization: London Health Sciences Centre (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14458
Record Dates: First submitted 2024-09-17; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Chronic Total Occlusion (CTO)
Keywords: CTO; Chronic Total Occlusion; Prehabilitation; Prehab; PCI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cardiac Prehabilitation for CTO Patients (Experimental): This single arm involves a 6-month cardiac pre-habilitation program designed for patients with chronic total occlusions (CTO) who are referred for percutaneous coronary intervention (PCI). Participants receive personalized cardiac rehabilitation, which includes physical exercise, medical optimization, and lifestyle modifications. The program aims to improve functional capacity and overall health before PCI. Assessments will be conducted at the start, after 6 months, and one month post-PCI if performed, with ongoing virtual follow-up for 5 months if PCI is not needed.
  Interventions: Other: Cardiac Prehabilitation Program

INTERVENTIONS:
Other: Cardiac Prehabilitation Program — Patients begin with a one-on-one assessment by a program cardiologist and a CR nurse, followed by a symptom-limited cardiopulmonary exercise test (CPET) to tailor their exercise regimen. The exercise program, based on the FITT (frequency, intensity, time, and type) principle, includes biweekly sessions either at home or at a commercial gym, with ongoing oversight by SJHC CRSP rehabilitation trainers. Additionally, participants have access to dietary counseling to optimize heart-healthy nutrition.

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility of a cardiac pre-hab program for patients with blocked arteries (CTO) who are referred for PCI treatment. The main questions it aims to answer are:

Can the pre-hab program improve patients' functional capacity before PCI? Does the pre-hab program impact the need for PCI based on improvements in patients' health?

Participants will:

Undergo an initial assessment including a physical exam, medication history, quality of life questionnaires, and blood work.

Complete a 6-month cardiac rehabilitation program. Have repeat assessments to evaluate improvements and determine if PCI is still needed.

If PCI is performed, be assessed again one month later for functional capacity improvements.

If PCI is not needed after 6 months, participants will be followed virtually for an additional 5 months.

DETAILED DESCRIPTION:
This is an investigator-initiated prospective single-arm single-center feasibility study of a cardiac pre-hab program for CTO patients referred for CTO PCI. All patients who undergo a coronary angiogram at the London Health Sciences Centre (LHSC) or who are referred to the LHSC CTO PCI program for the CTO PCI procedure within 1 year, will be screened for enrolment. Those who consent to participate in the trial will be referred to the Cardiac Rehabilitation and Secondary Prevention (CRSP) program for a period of cardiac rehabilitation (CR) prior to performing CTO PCI procedure (termed 'pre-hab'). Physical exam, prior history of medications, quality of life questionnaires and blood work will be performed at baseline during their initial pre-hab clinic consultation (Assessment 1). 6 months of pre-hab and medical optimization will be then initiated. After 6 months at Assessment 2 a repeat MIBI and functional Capacity will be reassessed and compare with baseline if there has been any improvement. Based on them, the need for CTO PCI will be redetermined. If CTO PCI is still indicated,(Assessment 3a) after one month of CTO-PCI will be performed to assess improvement in functional capacity.

On the other hand, if CTO-PCI is not required after 6 months the participant will be followed virtually by Cardiac Rehab for 5 months. A final Assessment 4 will be made at 6 month in both instances

ELIGIBILITY:
Inclusion Criteria:

1. The presence of a chronic total occlusion in at least one major coronary artery (diameter ≥ 2.5mm).
2. Patients who have an indication for percutaneous coronary intervention of a CTO, which includes the presence of:

   1. Angina or anginal-equivalent symptoms and
   2. Ischemia or viability in the CTO territory
3. Patient aged ≥18 years of age.

Exclusion Criteria:

1. Inability or refusal to participate in the study's cardiac rehabilitation program.
2. Participation in CR program in the last 1 year.
3. Life expectancy of < 12 months due to non-cardiovascular comorbidities.
4. Anatomy deemed unsuitable for CTO PCI.
5. Severe left main disease (angiographic stenosis ≥50%; fractional flow reserve ≤0.80; minimal lumen area <6mm2).
6. Severe valvular disease or valvular disease likely to require surgery or percutaneous valve replacement during the study period.
7. Pregnancy.
8. Acute coronary syndrome within two months.
9. Canadian Cardiovascular Society Class ≥III angina of recent onset.
10. Angina of any class with a rapidly accelerating pattern.
11. Cardiac transplant recipient.
12. Inability to understand the questionnaires used in the study.
13. Patients unable to provide consent for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the Prehab-CTO PCI program | 2 years
  Assessment of eligibility and recruitment rates using a traffic light system (green: feasible, Amber: feasible with modifications, Red: not feasible).
  Unit of measure: N/A (qualitative assessment)

SECONDARY OUTCOMES:
Effectiveness of the Prehab-CTO PCI Program | 2 years
  Assessment of changes in quality of life, exercise capacity, symptomatology, and depression scores at three time points: after the pre-hab program, after CTO PCI, and at 6 month follow-up. Durability of benefits will also be evaluated.
  Units of measure:
  Exercise Capacity: Distance in meters from the 6-Minute Walk Test (A longer distance indicates better exercise capacity, so higher values are associated with better outcomes.)
Effectiveness of the Prehab-CTO PCI Program | 2 years
  Assessment of changes in quality of life, exercise capacity, symptomatology, and depression scores at three time points: after the pre-hab program, after CTO PCI, and at 6 month follow-up. Durability of benefits will also be evaluated.
  Units of measure:
  Symptomatology: Seattle Angina Questionnaire score (0-100) with 100 representing the absence of angina and optimal physical function and quality of life related to angina.
Effectiveness of the Prehab-CTO PCI Program | 2 years
  Assessment of changes in quality of life, exercise capacity, symptomatology, and depression scores at three time points: after the pre-hab program, after CTO PCI, and at 6 month follow-up. Durability of benefits will also be evaluated.
  Units of measure:
  Depression: PHQ-9 score (0-24) a score from 0 to 24 is produced. Scores of 5, 10, 15 and 20 represent cutpoints for mild, moderate, moderately, and severe depression respectively.
Effectiveness of the Prehab-CTO PCI Program | 2 years
  Assessment of changes in quality of life, exercise capacity, symptomatology, and depression scores at three time points: after the pre-hab program, after CTO PCI, and at 6 month follow-up. Durability of benefits will also be evaluated.
  Units of measure:
  Quality of life: EQ-5D score (scale 0-1) 1 represents full health, 0 represents a health state equivalent to death.
Estimate of the incidence of cardiovascular events in CTO patients undergoing prehab | 2 years
  Estimation of the total number of cardiovascular events (including all-cause death, cardiovascular death, stroke, non-fatal myocardial infraction, hospitalization for cardiovascular causes, and unplanned revascularization) occuring during the prehab program.
  Unit of measure: estimate/count of events

CONTACTS AND LOCATIONS:
Overall Officials: Luiz F Ybarra, MD PhD MBA FRCPC, Principal Investigator — London Health Sciences Centre
Locations (1):
- University Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Not part of the study plan/design.

REFERENCES:
- [Background] Ybarra LF, Dautov R, Gibrat C, Dandona S, Rinfret S. Midterm Angina-Related Quality of Life Benefits After Percutaneous Coronary Intervention of Chronic Total Occlusions. Can J Cardiol. 2017 Dec;33(12):1668-1674. doi: 10.1016/j.cjca.2017.08.008. Epub 2017 Aug 19. PMID 29066329
- [Background] Ybarra LF, Rinfret S, Brilakis ES, Karmpaliotis D, Azzalini L, Grantham JA, Kandzari DE, Mashayekhi K, Spratt JC, Wijeysundera HC, Ali ZA, Buller CE, Carlino M, Cohen DJ, Cutlip DE, De Martini T, Di Mario C, Farb A, Finn AV, Galassi AR, Gibson CM, Hanratty C, Hill JM, Jaffer FA, Krucoff MW, Lombardi WL, Maehara A, Magee PFA, Mehran R, Moses JW, Nicholson WJ, Onuma Y, Sianos G, Sumitsuji S, Tsuchikane E, Virmani R, Walsh SJ, Werner GS, Yamane M, Stone GW, Rinfret S, Stone GW; Chronic Total Occlusion Academic Research Consortium. Definitions and Clinical Trial Design Principles for Coronary Artery Chronic Total Occlusion Therapies: CTO-ARC Consensus Recommendations. Circulation. 2021 Feb 2;143(5):479-500. doi: 10.1161/CIRCULATIONAHA.120.046754. Epub 2021 Feb 1. PMID 33523728